CLINICAL TRIAL: NCT04210271
Title: Testing an Intervention to Increase HIV Self-Testing Among Young, Black MSM
Acronym: TRUST
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: New York Blood Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 648283
Record Dates: First submitted 2018-01-29; First posted 2019-12-24 (Actual); Last update posted 2019-12-24 (Actual); Status verified 2019-12

CONDITIONS: HIV Testing

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- HIV Self-testing (Experimental): brief intervention to teach and support consistent self-testing with a friend
  Interventions: Behavioral: Buddy self-testing condition
- Generic Self-screening (Active Comparator): time and attention control providing basic self-screening education on a range of health outcomes
  Interventions: Behavioral: Control self-screening condition

INTERVENTIONS:
Behavioral: Buddy self-testing condition
  Arms: HIV Self-testing
Behavioral: Control self-screening condition
  Arms: Generic Self-screening

SUMMARY:
The investigators propose a study to design and test a brief intervention to increase uptake of consistent HIV self-testing among YBMSM using a novel and culturally-relevant "buddy system" approach. In the model, peer educators train pairs of YBMSM (or "buddies") to initiate self-testing and support each other in consistent self-testing (past 3 months) and sexual and AOD use risk reduction.

The specific aims of this developmental R01 study are:

1. To conduct qualitative formative research to adapt couples testing for self-testing with a buddy;
2. To assess the preliminary efficacy of the intervention to increase the proportion of YBMSM who self-test regularly over 12 months using a 2-arm randomized, controlled study design.

DETAILED DESCRIPTION:
Increasing HIV testing rates among young, Black men who have sex with men (YBMSM) is critical to reducing the disproportionate disease burden in the Black community. MSM comprised almost two-thirds of new HIV diagnoses in the United States (US) in 2010. We propose a study to design and test a brief intervention to increase uptake of consistent HIV self-testing among YBMSM using a novel and culturally-relevant "buddy system" approach. In our model, peer educators train pairs of YBMSM (or "buddies") to initiate self-testing and support each other in consistent self-testing (past 3 months) and sexual and AOD use risk reduction. We propose a study to design and test a brief intervention to increase uptake of consistent HIV self-testing among YBMSM using a novel and culturally-relevant "buddy system" approach. In the model, peer educators train pairs of YBMSM (or "buddies") to initiate self-testing and support each other in consistent self-testing (past 3 months) and sexual and AOD use risk reduction.

The specific aims of this developmental R01 study are:

1. To conduct qualitative formative research to adapt couples testing for self-testing with a buddy;
2. To assess the preliminary efficacy of the intervention to increase the proportion of YBMSM who self-test regularly (i.e., past three months) over 12 months using a 2-arm randomized, controlled study design.

The investigators will achieve the aims of the study in three phases, recruiting YBMSM using web- and app-based approaches. In Phase 1, the investigators conducted 30 in-depth interviews to identify barriers to, facilitators of, perceptions of and preferences for regular HIV self-testing, describe how AOD use and sexual behavior influence HIV self-testing behaviors, and assess participant perspectives on the proposed buddy intervention. In Phase 2, based on the formative research, the investigators adapted couples testing, integrating enhanced motivational interviewing techniques to create a brief, peer educator-delivered, face-to-face intervention. In Phase 3, for which the investigators currently seek IRB approval, the investigators will use web- and app-based, face-to-face and word-of-mouth approaches to recruit 376 HIV-negative, BMSM aged 18 to 34 who will be randomized as pairs to either the intervention arm (HIV testing together, HIV self-testing screening information and skills training; free test kits on demand; tailored booster messages) or the control arm (HIV testing separately, generic health screening information; free test kits on demand) and followed for 12 months to estimate the intervention's efficacy in increasing regular HIV self-testing according to self-report. If demonstrated to be efficacious, this innovative and efficient approach can be adapted easily for widespread distribution, with the potential to diffuse along naturally occurring, social networks among YBMSM.

ELIGIBILITY:
Inclusion Criteria:

* biological male at birth
* between 18 and 34 years of age
* self-identify Black, African American, Caribbean Black, African Black, multiethnic Black OR Latino/Hispanic
* reside in the NYC metropolitan area
* not HIV-infected (self-report)
* report insertive or receptive anal intercourse with another man in the past year
* ability to communicate in English
* provide informed consent for the study.
* willing to participate in the study with a friend or buddy.

Exclusion Criteria:

* currently enrolled in any other HIV research study involving HIV testing or an HIV vaccine trial

Ages: 18 Years to 34 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 402 (Actual)
Dates: Start 2016-06 (Actual); Primary Completion 2018-12 (Actual); Study Completion 2018-12 (Actual)

PRIMARY OUTCOMES:
Consistent HIV self-testing | 12 months
  One or more HIV self-test in past three months
Consistent HIV testing | 12 months
  One or more HIV test (any type) in past three months

REFERENCES:
- [Derived] Frye V, Nandi V, Paige MQ, McCrossin J, Lucy D, Gwadz M, Sullivan PS, Hoover DR, Wilton L; TRUST Study Team. TRUST: Assessing the Efficacy of an Intervention to Increase HIV Self-Testing Among Young Black Men Who have Sex with Men (MSM) and Transwomen. AIDS Behav. 2021 Apr;25(4):1219-1235. doi: 10.1007/s10461-020-03091-x. Epub 2020 Nov 15. PMID 33190178